CLINICAL TRIAL: NCT06968741
Title: Study to Assess the Safety and Effectiveness of the UrOActive® Artificial Urinary sPHincter In the treAtment of Stress Urinary Incontinence in Men
Brief Title: A Study to Assess the Safety and Effectiveness of the UrOActive® Artificial Urinary sPHincter (AUS)
Acronym: SOPHIA2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UroMems SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP CSO2307120900
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: Stress urinary incontinence; Artificial urinary sphincters
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Urinary Sphincter, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- UroActive AUS Implant (Experimental): Enrolled subjects who meet study eligibility criteria will proceed to receive the UroActive Artificial Urinary Sphincter (AUS) device
  Interventions: Device: Artificial Urinary Sphincter (AUS)

INTERVENTIONS:
Device: Artificial Urinary Sphincter (AUS) — AUS implant

SUMMARY:
Prospective, multicenter, single-arm study

ELIGIBILITY:
Key Inclusion Criteria:

* Male subjects aged ≥ 22 years old
* Able to read, comprehend and willing to sign an informed consent form
* Primary diagnosis of stress urinary incontinence for at least 6 months, as assessed by the investigator
* Appropriate surgical candidate with no medical or mental condition that would interfere with study procedures or confound study outcomes as assessed by the investigator

Key Exclusion Criteria:

* Currently enrolled or plans to enroll in another investigational device or clinical drug trial or has completed an investigational study (for urinary incontinence) in the past 3 months prior to informed consent
* Poor candidate for surgical procedures and/or anesthesia, as determined by investigator
* Currently implanted with an Active Implantable Medical Device (AIMD)
* Symptoms or diagnosis of urge incontinence or mixed incontinence (MI) with a predominant urgency component, as assessed by the investigator

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Responder rate at 26 weeks post-activation | 26 weeks
  Proportion of subjects who report greater than or equal to 50% reduction in the 24 hour Pad Weight Test (PWT) at 26 weeks compared with Baseline

OTHER OUTCOMES:
Proportion of subjects reporting change in overall impression of improvement (PGI-I) | 26 weeks
  Proportion of subjects reporting change in their overall impression of improvement with the use of their treatment as compared with Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — UroMems SAS
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No